CLINICAL TRIAL: NCT04384926
Title: Outcomes of Elective Cancer Surgery During the COVID-19 Pandemic Crisis: an International, Multicentre, Observational Cohort Study (CovidSurg-Cancer)
Brief Title: Outcomes of Elective Cancer Surgery During the COVID-19 Pandemic Crisis
Acronym: CovidSurg-Can
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: CSC-20200324
Record Dates: First submitted 2020-05-11; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Coronavirus; Cancer; Surgery
Keywords: Elective; Cancer Surgery
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Adult patients (aged ≥18 years), planned for curative cancer surgery, that have surgery completed during the COVID-19 pandemic
  Interventions: Procedure: Elective Cancer Surgery
- Cohort 2: Adult patients (aged ≥18 years), planned for curative cancer surgery, that have surgery delayed or cancelled during the COVID-19 pandemic
  Interventions: Procedure: Elective Cancer Surgery

INTERVENTIONS:
Procedure: Elective Cancer Surgery — Planned, curative cancer surgery

SUMMARY:
CovidSurg-Cancer is an international, multicentre, observational cohort study designed to evaluate the 30-day COVID-19 infection rates in elective cancer surgery during the COVID-19 pandemic.

Centres can elect to include one or more cancer types in the study, in any combination, depending on local expertise and capacity. During the pilot study, investigators should enrol patients with confirmed diagnoses of:

* Colorectal cancer
* Oesophagogastric cancer

As a rapid response study to the COVID-19 pandemic, included cancer types will evolve throughout the course of the CovidSurg-Cancer study period, for example, to include breast, liver, pancreatic, gynaecological, urological cancers, or sarcomas.

DETAILED DESCRIPTION:
The rapid emergence of the COVID-19 virus has led to a global impact on elective surgical care.

We have very little evidence to guide us. The magnitude and effects of these changes are uncertain. The safety of operating on patients electively with the risks of COVID-19 postoperative pneumonia is unknown.

High-quality data will allow policy planning at regional and hospital level for both this outbreak and future pandemics. CovidSurg-Cancer will run in parallel to CovidSurg (which is capturing outcomes of patients undergoing surgery for all indications with concurrent COVID-19).

The primary aim is to evaluate the 30-day COVID-19 infection rates in elective cancer surgery during the COVID-19 pandemic.

Secondary aims include; comparison of the 30-day postoperative mortality rate in cancer surgery patients that develop COVID-19 infection versus those who do not; an exploration of the scale of resource constraints related to the COVID-19 pandemic, and their impact on outcomes of elective cancer surgery; to explore variation in the selection of patients for continuing elective cancer surgery during the COVID-19 pandemic; to evaluate the impact of the COVID-19 pandemic on treatment pathways for cancers with a decision for surgical resection with curative intent.

This investigator-led, non-commercial, non-interventional study is extremely low to zero risk. This study does not collect any patient identifiable information and data will not be analysed at hospital-level.

ELIGIBILITY:
Centre Inclusion Criteria:

- Any centre performing elective cancer surgery

Inclusion Criteria (patient):

* Adults (age ≥18 years) with a confirmed diagnosis of an included cancer type
* Decision made for surgical management with a curative intent

Exclusion Criteria:

* Surgery planned with non-curative intent
* Planned neoadjuvant therapy without a firm date for surgery, or awaiting restaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients planned for curative cancer surgery that have surgery completed during the COVID-19 pandemic
  * Patients planned for curative cancer surgery that have surgery delayed or cancelled during the COVID-19 pandemic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day postoperative COVID-19 infection rate | 30 days
  Frequency of COVID-19 infection within 30 days

SECONDARY OUTCOMES:
30-day postoperative mortality rate | 30-days
  Number of deaths at 30-days post surgery
Postoperative critical care utilisation rate in high-risk cancer surgery patients. | 30-days
  Critical care utilisation in high-risk cancer surgery patients
Proportion of patients with delay of greater than 4 weeks from decision for surgery to date of surgery | More than 4 weeks from decision date
  Number of patients with a delay of more than 4 weeks from the decision taken for surgery to the date of surgery
Proportion of non-operated patients with progression to incurable disease by 3-months after decision for surgery | Up to 3-months
  Number of non-operated patients with progression to incurable disease by 3-months after decision for surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aneel Bhangu, Principal Investigator — University of Birmingham
Locations (1):
- Hospital del Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers

REFERENCES:
- [Derived] NIHR Global Health Research Unit on Global Surgery; STARSurg Collaborative. A prognostic model for use before elective surgery to estimate the risk of postoperative pulmonary complications (GSU-Pulmonary Score): a development and validation study in three international cohorts. Lancet Digit Health. 2024 Jul;6(7):e507-e519. doi: 10.1016/S2589-7500(24)00065-7. PMID 38906616
- [Derived] COVIDSurg Collaborative. Effect of COVID-19 pandemic lockdowns on planned cancer surgery for 15 tumour types in 61 countries: an international, prospective, cohort study. Lancet Oncol. 2021 Nov;22(11):1507-1517. doi: 10.1016/S1470-2045(21)00493-9. Epub 2021 Oct 5. PMID 34624250
- [Derived] Glasbey JC, Nepogodiev D, Simoes JFF, Omar O, Li E, Venn ML, Pgdme, Abou Chaar MK, Capizzi V, Chaudhry D, Desai A, Edwards JG, Evans JP, Fiore M, Videria JF, Ford SJ, Ganly I, Griffiths EA, Gujjuri RR, Kolias AG, Kaafarani HMA, Minaya-Bravo A, McKay SC, Mohan HM, Roberts KJ, San Miguel-Mendez C, Pockney P, Shaw R, Smart NJ, Stewart GD, Sundar Mrcog S, Vidya R, Bhangu AA; COVIDSurg Collaborative. Elective Cancer Surgery in COVID-19-Free Surgical Pathways During the SARS-CoV-2 Pandemic: An International, Multicenter, Comparative Cohort Study. J Clin Oncol. 2021 Jan 1;39(1):66-78. doi: 10.1200/JCO.20.01933. Epub 2020 Oct 6. PMID 33021869